CLINICAL TRIAL: NCT00091611
Title: Phase II Study in Metastatic Renal Cell Cancer Using Cultured, Tumor-Reactive Lymphocytes and Interleukin-2
Brief Title: Cultured White Cells Plus Interleukin-2 to Treat Advanced Kidney Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated due to low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040277; 04-C-0277; NCT00093574 (obsolete NCT alias)
Record Dates: First submitted 2004-09-11; First posted 2004-09-13 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Kidney Neoplasms
Keywords: Clinical Response; Intravenous; Intra-Arterial; Lymphodepletion; Traffic of Cells; T-Cell Transfer; Renal Cell Carcinoma; Metastatic Renal Cell Cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interleukin-2; Muromonab-CD3; Cyclophosphamide; fludarabine; Mesna

INTERVENTIONS:
Drug: IL-2 (interleukin-2)
Drug: OKT3
Drug: Cyclophosphamide
Drug: Fludarabine
Drug: Mesna

SUMMARY:
Background:

* Some patients with advanced kidney cancer have immune cells that can recognize and kill their cancer, but the cells are not active enough or numerous enough to accomplish this on their own.
* In recent studies of patients with advanced melanoma, some patients given special tumor-fighting cells (cells taken from the patient's tumor cells and grown in the laboratory) showed some anti-tumor response.

Objectives:

-To determine whether special tumor-fighting cells taken from the patient's blood or tumor and grown in the laboratory can cause tumors in patients with kidney cancer to shrink when they are given back to the patient along with interleukin-2.

Eligibility: Patients 18 years of age or older with advanced kidney cancer.

Design:

* Up to 29 patients will be treated in this study.
* Patients undergo tumor biopsy to collect tumor cells for creating special tumor-fighting cells for later infusion.
* Patients undergo apheresis to collect stem cells for later re-infusion. For apheresis, whole blood is collected through a needle in an arm vein and circulated through a cell-separating machine where the stem cells are extracted. The rest of the blood is returned through the same needle or a needle in the other arm.
* Before receiving the treated white cells, patients are given two drugs to suppress the immune system so the treated cells can work without interference from immune system cells. They are given cyclophosphamide over 2 days through a catheter (plastic tube inserted into a vein in the arm or neck) and fludarabine through the catheter over 15-30 minutes for the next 5 days.
* The day after the last dose of fludarabine, the tumor-fighting cells are infused through a vein over 10-20 minutes.
* Following the cell infusion, patients start treatment with high-dose interleukin-2 every 8 hours for a maximum of 12 doses.
* Patients are evaluated with x-ray studies about 1 month after receiving the cells and interleukin 2 (IL-2) to look for tumor response to treatment. Those who show significant improvement continue to receive treatment until the treated cells are used up or the patient no longer benefits or develops unacceptable side effects.

DETAILED DESCRIPTION:
Background:

One area of therapeutic advancement in immunotherapy has been to identify autologous tumor-reactive T-cells and expand them in vitro, and administer them in adoptive transfer back to patients. These T-cells have been obtained either from tumor infiltrating lymphocytes (TIL) which appear enriched for tumor-reactive T-cells or by in vitro stimulation of peripheral blood T-cells from cancer patients. Recent success in patients with melanoma has in large part been due to a T-cell expansion protocol described by Riddell et al. using anti-CD3 (cluster of differentiation 3) and irradiated allogeneic feeder cells and the use of conditioning chemotherapy prior to cell transfer. This current study uses the results of these Surgery Branch adoptive cell therapy trials to study their potential in patients with metastatic renal cell cancer.

Objectives:

The primary objective will be to determine whether adoptive lymphocyte transfer in conjunction with preparative lympho-depletion chemotherapy and interleukin-2 (IL-2) may result in clinical tumor regression in patients with metastatic renal cancer.

Eligibility:

Patients with metastatic renal cell cancer who have failed conventional therapy with interleukin-2, from whom tumor-reactive lymphocytes (from either peripheral blood, lymph nodes or tumor-infiltrating lymphocytes) can be obtained and expanded in vitro.

Patients must meet specific safety laboratory criteria, be able to tolerate interleukin 2 (IL-2), and have no concurrent major medical illnesses or symptomatic brain metastases.

Design:

All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day intravenous (IV)) on days -7 and -6 and fludarabine (25 mg/m^2/day intravenous (IV)) on days -5 through -1. On day 0 patients will receive an infusion of their own tumor-reactive T cells grown in vitro (greater than or equal to 5x10^8 cells for a cycle) and then begin high-dose IL-2 (720,000 IU/kg intravenous (IV) every 8 hours for up to 15 doses).

Clinical and Immunologic response will be evaluated about 3 to 5 weeks after the treatment regimen.

This trial will be conducted as a phase II trial using a two-stage MinMax design which will try to determine whether intravenous (IV) cell administration can produce a modest response rate targeted to be greater than or equal to 35 % (p1=0.35) as opposed to an undesirably low response rate of less than 15% (p0=0.15). If at least 3 patients of 15 have an objective response (partial response (PR) or complete response (CR)) accrual will proceed to 28 patients, with a projected accrual over three years.

ELIGIBILITY:
* INCLUSION CRITERIA: CELL HARVEST:
* Patients must have metastatic renal cell cancer.
* age greater than or equal to 18 years.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1 at entry to the trial.
* Life expectancy of greater than three months.
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are human immunodeficiency virus (HIV) seropositive can have decreased immune competence and can thus be less responsive to the experimental treatment and more susceptible to it's toxicities.)
* Seronegative for hepatitis B antigen.
* Seropositive for Epstein-Barr Virus (EBV).
* Patients with electrocardiogram (EKG) abnormalities, symptoms of cardiac ischemia or arrythmias or age greater than 50 years must have a normal stress cardiac test (stress thallium, stress multi-gated acquisition scan (MUGA), dobutamine echocardiogram or other stress test).
* Patients who have a recent prolonged history of cigarette smoking or symptoms of respiratory dysfunction must have pulmonary function testing with an forced expiratory volume in 1 second (FEV(1)) greater than 60% predicted.

EXCLUSION CRITERIA: CELL HARVEST:

-Active systemic infections, coagulation disorders, contra-indications to receiving interleukin-2 (IL-2) or major medical illnesses of the cardiovascular, respiratory or immune system.

INCLUSION CRITERIA: CELL INFUSION:

* Patients must have measurable metastatic renal cell cancer and have tumor progression after therapy with interleukin-2 (IL-2).
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1 at entry to the treatment phase of this trial.
* Platelet count greater than 100,000/mm^3.
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than three times the upper limit of normal.
* Serum creatinine less than or equal to 1.6 mg/dl.
* Total bilirubin less than or equal to 1.6 mg/dl or direct bilirubin less than or equal to 0.5 mg/dl.
* Life expectancy of greater than three months.
* At the time of T-cell transfer, the patient must have a T-cell population which has met the attached Certificate of Analysis for tumor recognition and safety testing.
* Any patient receiving interleukin-2 (IL-2) must sign a durable power of attorney.
* Male and Female patients must be willing to practice contraception during the treatment phase of this study..
* Patients with asymptomatic brain metastases may be considered eligible.

EXCLUSION CRITERIA: CELL INFUSION:

* Potentially effective therapy for renal cell cancer (RCC) within four weeks of the time the patient receives T-cell transfer (with the exception of local irradiation to non-evaluated sites).
* Requirement for steroid therapy.
* Active systemic infections, coagulation disorders, contra-indications to receiving interleukin-2 (IL-2) or major medical illnesses or the cardiovascular, respiratory or immune system.
* Pregnant patients and nursing mothers will be excluded because of the unknown effects of this therapy on the fetus or nursing infant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Determine whether Adoptive Lymphocyte Transfer in Conjunction with Preparative Lympho-depletion Chemotherapy and Interleukin-2 (IL-2) May result in Clinical Tumor Regression in Metastatic Renal Cancer

CONTACTS AND LOCATIONS:
Overall Officials: James Yang, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenberg SA, Zhai Y, Yang JC, Schwartzentruber DJ, Hwu P, Marincola FM, Topalian SL, Restifo NP, Seipp CA, Einhorn JH, Roberts B, White DE. Immunizing patients with metastatic melanoma using recombinant adenoviruses encoding MART-1 or gp100 melanoma antigens. J Natl Cancer Inst. 1998 Dec 16;90(24):1894-900. doi: 10.1093/jnci/90.24.1894. PMID 9862627
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2004-C-0277.html